CLINICAL TRIAL: NCT05474339
Title: The Effects of Cardiac Rehabilitation on Sleep Quality and Sleep Duration in Patients After Coronary Artery Bypass Graft: A Randomized Control Trial
Brief Title: The Effects of Cardiac Rehabilitation on Sleep Quality and Sleep Duration in Patients After Coronary Artery Bypass Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsien-Chum Wang, Physical therapy, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220504R
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft; Sleep Quality; Cardiac Rehabilitation
Keywords: Coronary Artery Disease; Coronary artery bypass graft; Sleep quality; Sleep duration; Cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Sleep Initiation and Maintenance Disorders | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac rehabilitation group (Experimental)
  Interventions: Other: Cardiac rehabilitation
- Control group (No Intervention)

INTERVENTIONS:
Other: Cardiac rehabilitation — Using Cardiac rehabilitation for patients after coronary artery bypass graft
  Arms: Cardiac rehabilitation group

SUMMARY:
This study aims to investigate the effects of cardiac rehabilitation on sleep quality and sleep duration in patients after coronary artery bypass graft.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is one of the common cardiovascular diseases, including myocardial infarction and unstable angina pectoris. Using the Global Burden of Disease statistical data analysis in 2020, Khan and other scholars found that the global prevalence of CAD is about 1,655 per 100,000 people, and the prevalence rate in Taiwan is about 1759 per 100,000 people, slightly higher than the global prevalence rate. Therefore, all countries in the world attach great importance to the prevention and treatment of CAD. In addition to common risk factors such as age, metabolic disease, smoking, and poor lifestyle habits such as insufficient physical activity, the literature indicates that sleep quality and sleep duration are also significantly associated with CAD. A 2011 meta-analysis by Francesco et al. pointed out that people who sleep less than 5 hours have a higher risk of CAD and are significantly associated with higher mortality rate. Patients with CAD who self-reported poor sleep quality and short sleep duration still had a high proportion after heart-related treatment. In 1993, Redeker tracked the related symptoms of patients after coronary artery bypass graft(CABG) and found that the sleep disturbance of patients did not improve, but increased. A systematic review of the literature by Liao et al. also found similar results. The sleep quality and sleep duration of patients after CABG can be improved over time, but a high proportion of patients still complain of sleep disturbance. Therefore, the influence of sleep disturbance in patients with CAD will persist, and studies have also suggested that persistent sleep disturbance will increase the readmission rate and mortality rate of patients with CAD. Therefore, it is very important to actively manage the sleep quality and sleep time of patients with CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-80 years old
* Have undergone CABG
* The score of PSQI > 5
* Can accomplish with instructions and complete the evaluation process
* Body mass index less than 35 Kg/m2

Exclusion Criteria:

* Diagnosed with
* Sleep apnea (e.g., obstructive sleep apnea, and central sleep apnea)
* Drug or alcohol dependence
* Psychology disease
* Neurological or musculoskeletal disorders that may interfere with CR
* Uncontrolled cardiac status (e.g., unstable angina, and uncontrolled arrhythmia)
* Women in pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change between baseline and 3 mons. after cardiac rehabilitation
  Range of 0-21, higher scores indicate worse sleep quality. Scores > 5 are taken to represent poor sleep quality
Actigraphy | Change between baseline and 3 mons. after cardiac rehabilitation
  Objective sleep parameter. Wear on the non-dominant wrist for 24 hrs. Can measure the total sleep time (TST), sleep onset latency (SOL), wake after sleep onset (WASO), sleep efficiency (SE)

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Change between baseline and 3 mons. after cardiac rehabilitation
  General level of daytime sleepiness . 8 self-rated questions. The chance of dozing is rated on a scale of 0-3. Range of 0-24, higher scores indicate worse daytime sleepiness. Scores > 10 are taken to represent excessive daytime sleepiness.
Visual analogue scale | Change between baseline and 3 mons. after cardiac rehabilitation
  Pain rating scales. Mark a 100 mm line to indicate pain intensity. 0 mm = no pain, 100 mm = worst pain
Hospital Anxiety and Depression Scale (HADS) | Change between baseline and 3 mons. after cardiac rehabilitation
  Range of 0-21, higher scores indicate worse anxiety or depression. Scores > 10 are taken to represent anxiety or depression
Cardiopulmonary exercise testing (CPET) | Change between baseline and 3 mons. after cardiac rehabilitation
  Gold standard for exercise capacity. Protocol: Starting form 0 watt, increase 10-15 watt/min. Test termination: Reach ≥ 85% of maximal HR, Respiratory exchange ratio (RER) > 1.10, Participants feel exhausted

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Chum Wang, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No